CLINICAL TRIAL: NCT06869161
Title: Comparison of the Effects of Stabilization Splint and Muscle Exercises on Pain and Muscle Thickness in Patients With Central Sensitization Caused by Myofascial Pain: A Randomized Controlled Clinical Trial
Brief Title: Comparison of Treatment Alternatives for Myofascial Pain Causing Central Sensitization
Acronym: Myofascialpain
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, İlke Çalışkan, Arş. Gör. Dt., Cukurova University
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Supportive Care
Other Study IDs: CU-PDT-IC-01
Record Dates: First submitted 2025-03-05; First posted 2025-03-11 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-03

CONDITIONS: Myofacial Pain; Central Sensitization
Keywords: central sensitization; myofacial pain; stabilization splints; muscle thickness; muscle exercises
MeSH Terms: conditions — Facial Pain | interventions — Exercise Therapy

STUDY DESIGN:
Intervention Model Description: Bilateral masseter and temporal muscle thicknesses of all participants will be measured and recorded with a Clarius L7 ultrasound device. Muscle thickness measurements will be repeated at week 2, week 4, week 8 of the treatments and pain report forms will be filled out. As of week 8, treatments will be terminated and patients will be called to the clinic for control visits at week 12 and muscle thickness measurements will be repeated and pain report forms will be filled.
Who Masked: Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control group (No Intervention): Participants were trained on the protection program.
- Stabilization splint group (Active Comparator): The participants will use occlusal splints that are digitally designed by transferring the measurements taken with intraoral scans (TRIOS5, 3Shape TRIOS A/S, Copenhagen, Denmark) to the exocad design program and produced by three-dimensional printers.
  Interventions: Device: Stabilization splint
- Exercises Group (Active Comparator): Participants will be given home-based exercise programs prepared by physical therapists.
  Interventions: Other: Muscle exercises
- Stabilization Splint and Exercises Group (Active Comparator): Participants will use occlusal splints, which are digitally designed by transferring the measurements taken with intraoral scans (TRIOS5, 3Shape TRIOS A/S, Copenhagen, Denmark) to the exocad design program and produced from 3D printers, and home exercise programs prepared by physical therapists will be given.
  Interventions: Device: Stabilization splint

INTERVENTIONS:
Device: Stabilization splint — Measurements will be taken from the patients with intraoral scans, transferred to the design program and a stabilization splint will be digitally designed. The designed splint will be produced from 3D printers.
  Other Names: exercises
  Arms: Stabilization Splint and Exercises Group; Stabilization splint group
Other: Muscle exercises — Muscle exercises prepared by physical therapists will be planned to relieve trigger points in the masticatory muscles.
  Arms: Exercises Group

SUMMARY:
Myofascial pain is a regional muscle pain condition characterized by hard local areas and tender bands, known for the presence of trigger points in muscle tissue. The treatment is to eliminate the etiologic factor. Regular exercise is recommended to relieve the trigger points. Occlusal splints, considered the gold standard in the treatment of temporomandibular joint disorders, are used to manage and control symptoms. In this study, patients between the ages of 18-45 years who applied to Çukurova University Faculty of Dentistry, Department of Prosthodontics with the complaint of myofascial pain and scored above 40 on the central sensitization scale will be taken as a sample.

DETAILED DESCRIPTION:
Patients scoring 40 and above on the CSI scale will be evaluated according to the Diagnostic Criteria - Diagnostic Criteria for Temporomandibular Disorders (DC-TMD) and four groups will be formed including the control group diagnosed with myofascial pain. Bilateral masseter and temporal muscle thicknesses of all participants will be measured and recorded with a Clarius L7 ( Vancouver, Canada) ultrasound device. The control group will be trained and asked to comply with the training until the study is completed. The participants in the first experimental group will use occlusal splints that are digitally designed by transferring the impressions taken with intraoral scanner (TRIOS5, 3Shape TRIOS A/S, Copenhagen, Denmark) to the exocad design program and printed on three-dimensional printers. Participants in the second experimental group will be given home-based exercise programs prepared by physical therapists. Participants in the third experimental group will use occlusal splints digitally designed by transferring the impressions taken with intraoral scans (TRIOS5, 3Shape TRIOS A/S, Copenhagen, Denmark) to the exocad design program and printed on three-dimensional printers and will be given home-based exercise programs prepared by physical therapists.

Muscle thickness measurements will be repeated at week 2, week 4, week 8 of the treatments and pain report forms will be filled out. As of week 8, treatments will be terminated and patients will be called to the clinic for control visits at week 12 and muscle thickness measurements will be repeated and pain report forms will be filled.

ELIGIBILITY:
Inclusion Criteria:

* Examination of bilateral masseter and temporal muscles for the presence of trigger points
* Score above 40 on the CSI scale

Exclusion Criteria:

* Noise during jaw movements (click, crepitation)
* Presence of systemic diseases involving joints (rheumatoid arthritis)
* Having received treatment for joint discomfort in the last six months (botox, splinting, exercise, counseling)
* Use of drugs affecting the central system (gabapentin, pregabalin, tricyclic antidepressants)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-05-12 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-25 (Estimated)

PRIMARY OUTCOMES:
Muscle Thickness | Baseline, 2 weeks, 4 weeks, 8 weeks, 12 weeks
  Bilateral masseter and temporal muscle thicknesses of the participants will be measured with an ultrasound device (Clarius L7, Vancouver, Canada) , muscle thickness differences will be evaluated and the time period in which the effectiveness of the treatments will be observed will be determined.

SECONDARY OUTCOMES:
Graded chronic pain scale | Baseline, 4 weeks, 8 weeks, 12 weeks
  A questionnaire (Graded Chronic Pain Scale -1 to 10 grades scale index-, will be used to assess changes in the amount and frequency of pain and its impact on daily life.

CONTACTS AND LOCATIONS:
Locations (1):
- Çukurova Üniversitesi Diş Hekimliği Fakültesi Protetik Diş Tedavisi Anabilim Dalı, Sarıçam, Balcalı Mahallesi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes